CLINICAL TRIAL: NCT04798352
Title: Follow-up Study in French Practice to Evaluate the Improvement of Gait and Pain Relief in Patients Treated With Endovascular Endovascular Treatment of de Novo Lesions of the Femoropopliteal Artery Above the Knee With LUTONIX®035 or RANGER TM Active Ballon
Brief Title: Follow-up Study in French Practice to Evaluate Improvements in Walking and Pain Relief in Patients Treated With Endovascular Treatment of de Novo Lesions of the Femoropopliteal Artery Above the Knee With LUTONIX®035 or RANGER TM Active Ballon
Acronym: EQUATEUR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire Dijon (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: STEINMETZ BOSTON BARD 2019
Record Dates: First submitted 2021-03-08; First posted 2021-03-15 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Drug-coated Balloon Catheter

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- LUTONIX(R)035 drug-coated balloon catheter (Experimental)
  Interventions: Other: 6-minute walk test; Other: WIQ functional questionnaire; Other: quality of life questionnaires (EQ5D5L and SF-36)
- RANGER TM drug-coated balloon catheter (Experimental)
  Interventions: Other: 6-minute walk test; Other: WIQ functional questionnaire; Other: quality of life questionnaires (EQ5D5L and SF-36)

INTERVENTIONS:
Other: 6-minute walk test — 6-minute walk test
Other: WIQ functional questionnaire — WIQ functional questionnaire
Other: quality of life questionnaires (EQ5D5L and SF-36) — quality of life questionnaires (EQ5D5L and SF-36)

SUMMARY:
This study is part of the subordination for the renewal of the registration of the LUTONIXR035 or RANGERTM drug coated balloon catheter by the CNEDiMTS following the transmission of the results of a French study on quality of life (evaluation of pain relief and walking evaluation criteria) for patients treated for de novo lesions of the femoropopliteal artery above the knee by endovascular treatment with LUTONIXR035 or RANGERTM drug-coated balloon catheters.

In accordance with the HAS practical guide on the approval of medical devices in France (November 2017), the protocol for this study was submitted in advance to the HAS and its suggestions were taken into account when drafting the objectives relative to the population to be included.

A second exhaustive study will be conducted in parallel using SNDS data to complete the CNEDiMTS application in order to evaluate, in the context of this registration renewal, the interest of the technique by documenting limb preservation, overall survival, the rate of re-interventions and the number of stents implanted.

ELIGIBILITY:
Inclusion Criteria:

* patient having given express oral consent
* patient to be treated by endovascular procedure with a LUTONIXR035 or RANGER TM drug coated balloon catheter according to the recommendations of the ANSM dated 13/05/2019 1 and possible updates of these recommendations.

Exclusion Criteria:

* pregnant or likely to be pregnant (a pregnancy test may be carried out if necessary according to the centre's practice)
* adult unable to express consent
* patient whose follow-up is considered impossible by the investigator (comprehension problem, planned move, ...)

Per-intervention exclusion criteria

* patient considered to have failed endovascular treatment (presence of residual stenosis of more than 30% after surgery despite the possible use of a stent.
* Patient operated on but for whom the balloon was not used during the procedure
* Patient operated but for whom another balloon than those under study was finally used during the operation

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 293 (Actual)
Dates: Start 2020-12-04 (Actual); Primary Completion 2026-01-08 (Actual); Study Completion 2026-01-08 (Actual)

PRIMARY OUTCOMES:
average score of the WIQ specific self-questionnaire | at inclusion
average score of the WIQ specific self-questionnaire | and at 12 months after surgery
  progression of the functional limitations for walking evaluated by the average score of the WIQ specific self-questionnaire 12 months after surgery

CONTACTS AND LOCATIONS:
Locations (1):
- Chu Dijon Bourgogne, Dijon, France